CLINICAL TRIAL: NCT03062358
Title: A Phase III Randomized Double-blind Study of Pembrolizumab Plus Best Supportive Care vs. Placebo Plus Best Supportive Care as Second-Line Therapy in Asian Subjects With Previously Systemically Treated Advanced Hepatocellular Carcinoma (KEYNOTE-394)
Brief Title: Study of Pembrolizumab (MK-3475) or Placebo Given With Best Supportive Care in Asian Participants With Previously Treated Advanced Hepatocellular Carcinoma (MK-3475-394/KEYNOTE-394)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-394; MK-3475-394 (Other: MSD)
Record Dates: First submitted 2017-02-21; First posted 2017-02-23 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD1; PD-1; PDL1; PD-L1; PDL2
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pembrolizumab + BSC (Experimental): Participants receive pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
  Interventions: Biological: pembrolizumab; Other: best supportive care (BSC)
- placebo + BSC (Placebo Comparator): Participants receive placebo by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
  Interventions: Drug: placebo; Other: best supportive care (BSC)

INTERVENTIONS:
Biological: pembrolizumab — Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®
  Arms: pembrolizumab + BSC
Drug: placebo — Normal saline solution administered as an IV infusion Q3W
  Arms: placebo + BSC
Other: best supportive care (BSC) — BSC will include pain management and management of other potential complications including ascites per local standards of care.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of pembrolizumab or placebo given with best supportive care (BSC) in Asian participants with previously systemically treated advanced hepatocellular carcinoma (HCC). The primary hypothesis of this study is that overall survival is prolonged in participants who receive pembrolizumab compared to those who receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has a HCC diagnosis confirmed by radiology, histology, or cytology (fibrolamellar, and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible)
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy and not amenable to a curative treatment approach.
* Has a Child-Pugh A liver score within 7 days prior to first dose of study medication
* Has a life expectancy of >3 months
* Has at least one measurable lesion based on RECIST version 1.1 as determined by investigator.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 7 days prior to receiving the first dose of study medication.
* Has documented objective radiographic progression during or after treatment with sorafenib or oxaliplatin-based chemotherapy, or else intolerance to sorafenib or oxaliplatin-based chemotherapy
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female and male participants of reproductive potential must agree to use adequate contraception starting from the first dose of study medication, throughout the study period, and for up to 120 days after the last dose of study medication

Exclusion Criteria:

* Is currently participating or has participated in a study with an investigational agent or using an investigational device within 4 weeks of the first dose of study medication
* Has received sorafenib or oxaliplatin-based chemotherapy within 14 days of first dose of study medication
* Has had esophageal or gastric variceal bleeding within the last 6 months
* Has clinically apparent ascites on physical examination
* Has portal vein invasion at the main portal branch (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months
* Has had a solid organ or hematologic transplant
* Has had prior systemic therapy for HCC in the advanced (incurable) setting other than sorafenib or oxaliplatin-based chemotherapy, prior to start of study medication
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has received locoregional therapy to liver (transcatheter chemoembolization [TACE], transcatheter embolization [TAE], hepatic arterial infusion [HAI], radiation, radioembolization, or ablation) within 4 weeks prior to the first dose of study medication
* Has had major surgery to liver or other site within 4 weeks prior to the first dose of study medication
* Has had a minor surgery ≤7 days prior to the first dose of study medication
* Has not recovered adequately (i.e., Grade ≤1 or baseline) from the toxicity and/or complications from any intervention prior to study start
* Has a diagnosed additional malignancy within 3 years prior to first dose of study medication with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cancers
* Has a known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Is pregnant or breast feeding or expecting to conceive or father starting from the first dose of study medication, throughout the study period, and for up to 120 days after the last dose of study medication
* Has received prior immunotherapy with an anti-Programmed Cell Death Receptor 1 (PD-1), Programmed Cell Death Receptor Ligand 1 (anti-PD-L1), or anti-Programmed Cell Death Receptor Ligand 2 (PD-L2) or has previously participated in clinical studies with pembrolizumab
* Has a known history of human immunodeficiency virus (HIV)
* Has untreated active Hepatitis B
* Has Hepatitis C in which participants received therapy for HCV <4 weeks prior to receiving pembrolizumab
* Has received a live vaccine within 30 days prior to the first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (41):
- China (28):
  - Anhui Provincial Hospital ( Site 0032), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0005), Hefei, Anhui
  - Fuzhou General Hospital of Nanjing Military Command ( Site 0019), Fuzhou, Fujian
  - The First People s Hospital of Foshan ( Site 0033), Foshan, Guangdong
  - Guangdong General Hospital ( Site 0015), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0007), Harbin, Heilongjiang
  - Wuhan Tongji Hospital ( Site 0021), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0035), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0027), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 0026), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 0003), Nanjing, Jiangsu
  - The 81st Hospital of PLA ( Site 0016), Nanjing, Jiangsu
  - Nantong Tumor Hospital ( Site 0028), Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University ( Site 0025), Suzhou, Jiangsu
  - Yangzhou No.1 People's Hospital ( Site 0023), Yangzhou, Jiangsu
  - Jilin Province Cancer Hospital, Department of Chemotherapy ( Site 0002), Changchun, Jilin
  - The First Hospital Of Jilin University ( Site 0001), Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University ( Site 0022), Dalian, Liaoning
  - Fudan University Shanghai Cancer Center ( Site 0024), Shanghai, Shanghai Municipality
  - The first affiliated Hospital of Xi an Jiaotong University ( Site 0014), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0030), Chengdu, Sichuan
  - The First affiliated Hospital Zhejing University ( Site 0034), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0011), Hangzhou, Zhejiang
  - Beijing Cancer Hospital ( Site 0010), Beijing
  - Bengbu Medical College First Affiliated Hospital ( Site 0020), Bengbu
  - The Second Affiliated Hospital of Anhui Medical University ( Site 0008), Hefei
  - Zhongshan Hospital Fudan University ( Site 0012), Shanghai
  - Renji Hosp,Shanghai Jiao Tong University School of Medicine ( Site 0017), Shanghai
- Hong Kong (3):
  - Hong Kong Sanatorium Hospital ( Site 0053), Hong Kong
  - Pamela Youde Nethersole Eastern Hospital ( Site 0052), Hong Kong
  - Princess Margaret Hospital. ( Site 0051), Hong Kong
- Malaysia (3):
  - University Malaya Medical Centre ( Site 0091), Kuala Lumpur, Kuala Lumpur
  - Beacon Hospital Sdn Bhd ( Site 0092), Petaling Jaya, Selangor
  - Hospital Universiti Kebangsaan Malaysia ( Site 0093), Cheras
- South Korea (4):
  - Seoul National University Hospital ( Site 0074), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0073), Seoul
  - Asan Medical Center ( Site 0072), Seoul
  - Samsung Medical Center ( Site 0071), Seoul
- Taiwan (3):
  - Chia-Yi Chang Gung Memorial Hospital ( Site 0133), Chiayi City
  - China Medical University Hospital ( Site 0131), Taichung
  - National Cheng Kung University Hospital ( Site 0132), Tainan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Qin S, Chen Z, Fang W, Ren Z, Xu R, Ryoo BY, Meng Z, Bai Y, Chen X, Liu X, Xiao J, Ho GF, Mao Y, Wang X, Ying J, Li J, Zhong W, Zhou Y, Siegel AB, Hao C. Pembrolizumab Versus Placebo as Second-Line Therapy in Patients From Asia With Advanced Hepatocellular Carcinoma: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2023 Mar 1;41(7):1434-1443. doi: 10.1200/JCO.22.00620. Epub 2022 Dec 1. PMID 36455168
- [Derived] Finn RS, Gu K, Chen X, Merle P, Lee KH, Bouattour M, Cao P, Wang W, Cheng AL, Zhu L, Lim HY, Kudo M, Pan Y, Chang TT, Edeline J, Li W, Yang P, Li C, Li J, Siegel AB, Qin S. Second-line pembrolizumab for advanced HCC: Meta-analysis of the phase III KEYNOTE-240 and KEYNOTE-394 studies. JHEP Rep. 2025 Feb 4;7(6):101350. doi: 10.1016/j.jhepr.2025.101350. eCollection 2025 Jun. PMID 40486134
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants at least 18 years of age with advanced hepatocellular carcinoma (HCC) after progression on or intolerance to sorafenib or oxaliplatin-based chemotherapy with no curative option were enrolled in this study.
Groups:
- Pembrolizumab + BSC: Participants received 200 mg pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus best supportive care (BSC).
- Placebo + BSC: Participants received placebo by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
Period: Overall Study
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Started (All randomized participants) | 300 | 153
Treated (First Course Pembrolizumab) | 299 | 153
Second Course (Second Course Pembrolizumab) | 12 | 0
Completed | 0 | 0
Not Completed | 300 | 153
Not completed — Death | 269 | 145
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Sponsor Decision | 29 | 7

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab + BSC: Participants received 200 mg pembrolizumab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + BSC | Placebo + BSC | Total
Number analyzed (Participants) | 300 | 153 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.1) | 52.0 (12.9) | 53.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 27 | 70
  Male | 257 | 126 | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 300 | 153 | 453
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 300 | 153 | 453
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Macrovascular Invasion [Count of Participants; unit: Participants] — Per Case Report Form
  Participants
    Yes | 33 | 17 | 50
    No | 267 | 136 | 403
Alpha-Fetoprotein (α-Fetoprotein) [Count of Participants; unit: Participants] — Per Lab
  Participants
    < 200 ng/mL | 131 | 75 | 206
    ≥ 200 ng/mL | 169 | 78 | 247
Region [Count of Participants; unit: Participants] — China comprises: China mainland, Hong Kong, and Taiwan; Ex-China comprises: South Korea and Malaysia.
  Participants
    China | 255 | 132 | 387
    Ex-China | 45 | 21 | 66

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to death due to any cause, based on the Kaplan-Meier method for censored data.
Time Frame: Up to approximately 4 years
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 300 | 153
Months | 14.6 [12.6 to 18.0] | 13.0 [10.5 to 15.1]
Statistical Analysis 1: Comparison: Pembrolizumab + BSC vs Placebo + BSC; Test type: Superiority; p = 0.0180, One-sided p-value — Log-rank test; Stratified by macrovascular invasion, α-Fetoprotein and region with all cells that correspond to macrovascular invasion=Yes combined; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.63 to 0.99] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Stratified by macrovascular invasion (Yes vs. No), α-Fetoprotein (ng/mL) (< 200 vs. ≥ 200) and region (China vs. ex-China) with all cells that correspond to macrovascular invasion=Yes combined

2. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is the time from randomization to first documented disease progression or death due to any cause per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) based on the Kaplan-Meier method for censored data.
Time Frame: Up to approximately 4 years
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 300 | 153
Months | 2.6 [1.5 to 2.8] | 2.3 [1.4 to 2.8]
Statistical Analysis 1: Comparison: Pembrolizumab + BSC vs Placebo + BSC; Test type: Superiority; p = 0.0032, One-sided p-value — Log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.92] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is the percentage of participants who achieve complete response (CR) or partial response (PR) with confirmation per RECIST 1.1 by BICR. CR is the disappearance of all target lesions; PR is at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Up to approximately 4 years
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 300 | 153
Percentage of participants | 12.7 [9.1 to 17.0] | 1.3 [0.2 to 4.6]
Statistical Analysis 1: Comparison: Pembrolizumab + BSC vs Placebo + BSC; Difference in % vs Placebo; Test type: Other; p = 0.00004, One-sided p-value for testing; H0: difference in % =0 versus H1: difference in % > 0; Percent Difference = 11.4, 95% CI 2-sided [6.7 to 16.0] — Difference in % vs Placebo; Based on Miettinen & Nurminen method stratified by macrovascular invasion (Yes vs. No), α-Fetoprotein (ng/mL) (< 200 vs. >= 200) and region (China vs. ex-China) with all cells that correspond to macrovascular invasion=Yes combined

4. Secondary Outcome: Duration Of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR is the time from first documented evidence of CR or PR per RECIST 1.1 by BICR until disease progression per RECIST 1.1 by BICR or death, based on Kaplan-Meier method for censored data. CR is the disappearance of all target lesions; PR is at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Up to approximately 4 years
Population: All randomized participants with CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 41 | 2
Months | 23.9 [2.6 to 44.4] | 5.6 [3.0 to 5.6]

5. Secondary Outcome: Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DCR is the percentage of participants who achieve CR, PR, or stable disease (SD) for ≥5 weeks prior to evidence of disease progression per RECIST 1.1 by BICR. CR is the disappearance of all target lesions; PR is at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Up to approximately 4 years
Population: All randomized participants based on the treatment group to which they were randomized, who achieved CR, PR, or SD for ≥5 weeks prior to evidence of disease progression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 158 | 73
Percentage of participants | 52.7 [46.8 to 58.4] | 47.7 [39.6 to 55.9]
Statistical Analysis 1: Comparison: Pembrolizumab + BSC vs Placebo + BSC; Difference in % vs Placebo; Test type: Other; p = 0.13281, One-sided p-value for testing; H0: difference in % =0 versus H1: difference in % > 0; Percent Difference = 5.4, 95% CI 2-sided [-4.1 to 14.8] — Difference in % vs Placebo; Based on Miettinen & Nurminen method stratified by macrovascular invasion (Yes vs. No), α-Fetoprotein (ng/mL) (< 200 vs. ≥ 200) and region (China vs. ex-China) with all cells that correspond to macrovascular invasion=Yes combined

6. Secondary Outcome: Time To Progression (TTP) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: TTP is the time from randomization to first documented disease progression per RECIST 1.1 by BICR, based on Kaplan-Meier method for censored data.
Time Frame: Up to approximately 4 years
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 300 | 153
Months | 2.7 [1.5 to 2.8] | 1.7 [1.4 to 2.8]
Statistical Analysis 1: Comparison: Pembrolizumab + BSC vs Placebo + BSC; Test type: Other; p = 0.0019, One-sided p-value — Log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.90] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy.
Time Frame: Up to approximately 30 months.
Population: Randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 299 | 153
Participants | 283 | 147

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 7
Time Frame: Up to approximately 27 months.
Population: Randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + BSC | Placebo + BSC
Number analyzed (Participants) | 299 | 153
Participants | 38 | 13

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization up to approximately 7 years. Adverse events: from first treatment up to approximately 7 years.
Description: All-cause mortality population: All randomized participants. Adverse events population: Randomized participants who received at least 1 dose of study intervention. The following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Groups:
- Pembrolizumab First Course: Participants received 200 mg pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
- Placebo First Course: Participants received placebo by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus BSC.
- Pembrolizumab Second Course: Eligible participants randomized to the pembrolizumab first course who stopped pembrolizumab with stable disease (SD) or better, initiated a second course of pembrolizumab at the investigator's discretion at 200 mg of each 3 week cycle for up to 17 cycles up to approximately an additional year
Arm/Group | Pembrolizumab First Course | Placebo First Course | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 263/300 | 146/153 | 8/12
Serious Adverse Events (participants affected / at risk) | 76/299 | 31/153 | 1/12
Other Adverse Events (participants affected / at risk) | 272/299 | 135/153 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=299) | Placebo First Course (N=153) | Pembrolizumab Second Course (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 11 (11) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B DNA increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=299) | Placebo First Course (N=153) | Pembrolizumab Second Course (N=12)
Anaemia (Blood and lymphatic system disorders) | 45 (55) | 16 (17) | 1 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 16 (16) | 3 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 29 (35) | 11 (13) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 17 (18) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 20 (26) | 12 (12) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 17 (20) | 4 (5) | 0 (0)
Ascites (Gastrointestinal disorders) | 15 (16) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 27 (29) | 10 (14) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 47 (76) | 14 (20) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (24) | 8 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (25) | 10 (11) | 0 (0)
Asthenia (General disorders) | 18 (22) | 11 (13) | 0 (0)
Fatigue (General disorders) | 19 (20) | 9 (10) | 0 (0)
Malaise (General disorders) | 12 (14) | 10 (10) | 0 (0)
Pyrexia (General disorders) | 53 (70) | 21 (34) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 14 (16) | 8 (8) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 32 (37) | 10 (12) | 0 (0)
Alanine aminotransferase increased (Investigations) | 90 (138) | 36 (47) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 107 (162) | 45 (59) | 5 (7)
Bilirubin conjugated increased (Investigations) | 20 (26) | 7 (7) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 43 (60) | 15 (19) | 2 (2)
Blood bilirubin increased (Investigations) | 83 (142) | 40 (48) | 1 (1)
Blood creatinine increased (Investigations) | 10 (13) | 4 (4) | 1 (1)
Blood glucose increased (Investigations) | 9 (13) | 3 (4) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 15 (18) | 5 (8) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 54 (62) | 23 (25) | 3 (3)
Hepatitis B DNA increased (Investigations) | 15 (25) | 5 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 30 (41) | 10 (11) | 0 (0)
Neutrophil count decreased (Investigations) | 41 (98) | 17 (25) | 0 (0)
Platelet count decreased (Investigations) | 65 (134) | 25 (34) | 0 (0)
Weight decreased (Investigations) | 24 (26) | 6 (6) | 0 (0)
White blood cell count decreased (Investigations) | 51 (128) | 21 (33) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 44 (50) | 14 (18) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (28) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 12 (19) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 36 (46) | 13 (14) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (24) | 8 (12) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (23) | 7 (8) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 17 (23) | 9 (12) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (28) | 9 (11) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 12 (16) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (20) | 4 (4) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 31 (33) | 10 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (44) | 13 (16) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 35 (49) | 6 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 44 (54) | 8 (8) | 0 (0)
Hypertension (Vascular disorders) | 18 (22) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (2):
  • Study Protocol (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03062358/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT03062358/SAP_001.pdf